CLINICAL TRIAL: NCT01000480
Title: Phase 2 Study of Pemetrexed and Cisplatin as Induction, Followed by Pemetrexed and Cisplatin With Concurrent Thoracic Radiotherapy, in Patients With Unresectable, Locally Advanced, Stage III, Nonsquamous Non-Small Cell Lung Cancer
Brief Title: A Study of Pemetrexed and Cisplatin, in Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13099; H3E-EW-S128 (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed (Experimental): Pemetrexed and cisplatin are given as induction therapy followed after by pemetrexed and cisplatin with concurrent radiotherapy.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Radiation: Thoracic Radiotherapy

INTERVENTIONS:
Drug: Pemetrexed — 500 milligrams per square meter (mg/m²) intravenous infusion on Day 1 of a 21 day cycle for 2 cycles: with possibility of 2 additional cycles.
  Other Names: Alimta; LY231514
Drug: Cisplatin — 75 mg/m² intravenous infusion on Day 1 of a 21 day cycle for 2 cycles; with the possibility of 2 additional cycles.
Radiation: Thoracic Radiotherapy — Administered at 2 gray (Gy)/fraction after completion of the pemetrexed and cisplatin infusions on Day 1 of Cycle 3 and will continue daily (5 days per week) until the total delivered dose reaches a therapeutic goal of 66 Gy, over approximately 7 weeks.

SUMMARY:
This trial investigates pemetrexed and cisplatin followed by pemetrexed and cisplatin in combination with radiotherapy in participants with locally advanced, non-small cell lung cancer (NSCLC). The purpose of the study is to assess the antitumor activity as measured by progression free survival 1 year after start of treatment with study drug.

DETAILED DESCRIPTION:
The participants will receive 2 cycles of pemetrexed and cisplatin. If the participants achieve complete response, partial response or stable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, have ≤35% of the total calculated lung volume receive more than 20 Gy (V20) according to the 3-dimensional (3-D) radiotherapy planning Dose Volume Histograms, have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, have no residual neurological toxicity > Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE), they will receive 2 additional cycles of pemetrexed and cisplatin, combined with radiotherapy. The combination of radiotherapy will begin 22 to 36 days after completion of the second infusion of induction therapy with pemetrexed-cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of unresectable nonsquamous Stage IIIA or Stage IIIB (without malignant pleural/pericardial effusions) NSCLC.
* Have an ECOG performance status of 0 or 1.
* Previous radiation therapy should have been limited and must not have included thoracic radiation, whole pelvis radiation, or radiation to >25% of the participant's bone marrow, participants must have recovered from the toxic effects of radiation treatment prior to study enrollment (except for alopecia). Prior radiotherapy must be completed 30 days before study entry.
* Have at least 1 unidimensionally measurable lesion meeting RECIST guidelines, version 1.0.
* Estimated life expectancy of at least 12 weeks.
* Participant compliance and geographic proximity that allow adequate follow-up.
* Adequate bone marrow reserve, hepatic-, renal- and pulmonary function.
* Participants must sign an Informed Consent Document.
* Participants must have a total lung V20 less than or equal to 35%.
* For women: Must be surgically sterile, postmenopausal, or compliant with a medically approved contraceptive regimen, during and for 6 months after the treatment period; must have a negative serum pregnancy test within 7 days before study enrollment and must not be breast-feeding. For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 6 months after the treatment period.
* Have not received prior systemic anticancer therapy for NSCLC.

Exclusion Criteria:

* Have received treatment within the last 30 days of enrollment with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have previously completed or withdrawn from this study or any other study investigating pemetrexed.
* Have a serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the participant's ability to adhere to the protocol.
* Have a serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV.
* Have had a prior malignancy other than NSCLC, carcinoma in situ of the cervix, or non-melanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence. Participants with a history of low-grade (Gleason score less than or equal to 6) localized prostate cancer will be eligible even if diagnosed less than 5 years previously.
* Are receiving concurrent administration of any other antitumor therapy.
* Have had weight loss of more than 10% over the previous 3 months before study entry.
* Are unable to interrupt aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose less than or equal to 1.3 grams per day, for at least 2 days before (5 days for long-acting agents), the day of, and for at least 2 days after administration of pemetrexed.
* Are unable or unwilling to take folic acid or vitamin B12 supplementation.
* Are unable or unwilling to take corticosteroids.
* Have received a recent yellow fever vaccination (within 30 days of enrollment) or are receiving concurrent yellow fever vaccination.
* Have known hypersensitivity to pemetrexed, cisplatin, or any of the excipients in these medicinal products.
* Have evidence of clinical hearing loss.
* Have clinically significant third-space fluid collections, that cannot be controlled by drainage or other procedures prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-10; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5 PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Mans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hemer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuremberg
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avellino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perugia
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study treatment had 2 phases and follow-up. Induction phase: 2 cycles of pemetrexed-cisplatin. Then, if eligible, the concurrent phase: 2 more cycles of pemetrexed-cisplatin and thoracic radiotherapy. Follow-up period: Started when treatment discontinued or completed, and lasted up to 2 years after first dose of pemetrexed.
Groups:
- Pemetrexed, Cisplatin, and Thoracic Radiotherapy: Induction phase (2 cycles). Pemetrexed: 500 milligrams per square meter (mg/m²) intravenous infusion on Day 1 of 21-day cycle. Cisplatin: 75 mg/m² intravenous infusion on Day 1 of 21-day cycle.
  Participants eligible for concurrent phase (2 more cycles of pemetrexed-cisplatin treatment and radiotherapy) if they had complete response, partial response, or stable disease (Response Evaluation Criteria in Solid Tumors guidelines), total lung volume receiving more than 20 gray (Gy) ≤35% (dose volume histogram), 0 or 1 Eastern Cooperative Oncology Group performance status, no residual neurological toxicity >Grade 2 (Common Terminology Criteria for Adverse Events).
  Thoracic Radiotherapy: 2 Gy/fraction after completion of pemetrexed and cisplatin infusions on Day 1 of Cycle 3 and continued daily (5 days per week) until total delivered dose was 66 Gy, over approximately 7 weeks.
  Folic acid, Vitamin B12 supplements, and prophylactic dexamethasone administered per approved pemetrexed label.
Period: Induction Phase
Arm/Group | Pemetrexed, Cisplatin, and Thoracic Radiotherapy
Started | 90
Received at Least 1 Dose of Either Drug | 90
Death (Any Cause) or Disease Progression | 8 (Participants who died (any cause) or had disease progression considered to have completed phase.)
Completed | 83
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Entry Criteria Not Met | 3
Period: Concurrent Therapy Phase
Arm/Group | Pemetrexed, Cisplatin, and Thoracic Radiotherapy
Started | 75 (Eight participants (pts) who completed Induction Phase, not eligible for Concurrent Therapy Phase.)
Death (Any Cause) or Disease Progression | 1 (Pts who died (any cause) or had disease progression considered to have completed the phase.)
Completed | 65
Not Completed | 10
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Period: Follow-Up Period
Arm/Group | Pemetrexed, Cisplatin, and Thoracic Radiotherapy
Started | 88 (One pt lost to follow-up during induction, 1 pt died in concurrent therapy, both not enter follow-up)
Completed | 88
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: participants who received at least 1 dose of study drug (pemetrexed or cisplatin).
Arm/Group | Pemetrexed, Cisplatin, and Thoracic Radiotherapy
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 51
Race/Ethnicity, Customized [Number; unit: participants]
  White | 90
Region of Enrollment [Number; unit: participants]
  France | 9
  Spain | 17
  Germany | 42
  Italy | 22
Stage of Disease [Number; unit: participants] — Classification based on American Joint Committee on Cancer (AJCC) Staging System for lung cancer (sixth edition, 2002). Disease stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage IIIA is a locally advanced cancer that spread to lymph nodes within the chest area. Stage IIIB is a locally advanced cancer that spread to nearby tissue or far away lymph nodes, or has fluid, containing cancer cells, built up between the layers lining the lungs.
  participants
    Stage IIIA | 32
    Stage IIIB | 56
    Stage IV | 2
Eastern Cooperative Oncology Group (ECOG) performance status (PS) [Number; unit: participants] — ECOG PS classified participants according to their functional impairment. Scores ranged from 0 (Fully Active) to 5 (Death). 0=Fully Active; 1=Ambulatory, Restricted Strenuous Activity; 2=Ambulatory, No Work Activities; 3=Partially Confined to Bed, Limited Self Care; 4=Completely Disabled; and 5=Death.
  participants
    ECOG PS=0 | 59
    ECOG PS=1 | 31
    ECOG PS=2 | 0
Initial pathological diagnosis [Number; unit: participants] — The number of participants with an initial pathological diagnosis of Adenocarcinoma (lung), Carcinoma (large cell, lung), Carcinoma [non-small cell, lung, not otherwise specified (NOS)], Carcinoma (non-small cell, lung, poorly differentiated).
  participants
    Adenocarcinoma (lung) | 81
    Carcinoma (large cell, lung) | 7
    Carcinoma (non-small cell, lung, NOS) | 1
    Carcinoma (non-small cell, poorly differentiated) | 1
Current Tobacco Use [Number; unit: participants]
  Never used tobacco | 7
  Former user of tobacco | 55
  Current use of tobacco | 28

OUTCOME MEASURES:

1. Primary Outcome: 1 Year Progression Free Survival
Description: Progression free survival (PFS) was defined as the time from study enrollment to the first observation of progressive disease (PD) or death from any cause. For participants not known to have died as of the data cut-off date and who did not have objective PD, PFS was censored at the date of the last objective progression-free disease assessment. For participants who received subsequent systemic anticancer therapy (after discontinuation from the study drug) prior to objectively determined PD or death, PFS was censored at the date of the last objective progression-free disease assessment prior to start of postdiscontinuation chemotherapy. If a participant did not have a complete baseline disease assessment, then PFS was censored at the enrollment date, regardless whether or not objectively determined PD or death had been observed for the participant.
Time Frame: Date of first dose to date of objectively determined PD or death [every cycle up to 4 cycles and then every 3 months up to 1 year (1 cycle=21 days)]
Population: Intent-to-treat population: participants who received at least 1 dose of either study drug (pemetrexed or cisplatin). The number of participants censored was 35.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed, Cisplatin, and Thoracic Radiotherapy
Number analyzed (Participants) | 90
percentage of participants | 53.7 [44.8 to 62.5]
Statistical Analysis 1: Comparison: Pemetrexed, Cisplatin, and Thoracic Radiotherapy; Null hypothesis (H0): 1-year PFS ≤45% and the alternative hypothesis (H1): 1-year PFS ≥60%, at a 2-sided alpha level of 5%, assuming that PFS time followed an exponential distribution; Test type: Superiority or Other; p = 0.0645, maximum likelihood estimate — P-value for H0 which compared the investigational regimen to historical data

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was the duration from enrollment to death due to any cause. Participants who were alive were censored at the last contact.
Time Frame: Date of first dose to date of death (up to 35.4 months)
Population: Intent-to-treat population: participants who received at least 1 dose of study drug (pemetrexed or cisplatin). The number of participants censored was 45.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed, Cisplatin, and Thoracic Radiotherapy
Number analyzed (Participants) | 90
months | 26.2 [16.7 to NA] — The upper 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

3. Secondary Outcome: Number of Participants With an Objective Tumor Response
Description: Participants with confirmed complete response (CR), confirmed partial response (PR), stable disease (SD), or progressive disease (PD) according to Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria, as well as participants with a not evaluable/tumor response unknown. CR: disappearance of all tumor lesions. PR: either a) at least a 30% decrease in sum of longest diameter (LD) of target lesions taking as a reference baseline sum LDs, or b) complete disappearance of target lesions, with persistence (not worsening) of 1 or more nontarget lesions. In either case, no new lesions appeared. SD: small changes that did not meet above criteria. PD: at least a 20% increase in sum of LD of target lesions taking as reference smallest sum LD recorded since treatment started or appearance of 1 or more new lesions. Participants who discontinued study treatment (for reasons other than progression) before entering concurrent phase were considered to have non-evaluable response.
Time Frame: Date of first dose through end of follow-up [up to 30 weeks (1 cycle=21 days)]
Population: Intent-to-treat population: Participants who received at least 1 dose of study drug (pemetrexed or cisplatin).
Measure: Number; unit: participants
Arm/Group | Pemetrexed, Cisplatin, and Thoracic Radiotherapy
Number analyzed (Participants) | 90
participants
  Complete Response | 9
  Partial Response | 45
  Stable Disease | 16
  Disease Progression | 12
  Not evaluable/Response unknown | 8

ADVERSE EVENTS:
Arm/Group | Pemetrexed, Cisplatin, and Thoracic Radiotherapy
Serious Adverse Events (participants affected / at risk) | 23/90
Other Adverse Events (participants affected / at risk) | 85/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed, Cisplatin, and Thoracic Radiotherapy (N=90)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) — Event resulted in death
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) — Event resulted in death
Radiation oesophagitis (Injury, poisoning and procedural complications) | 8 (9)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed, Cisplatin, and Thoracic Radiotherapy (N=90)
Anaemia (Blood and lymphatic system disorders) | 7 (8)
Leukopenia (Blood and lymphatic system disorders) | 12 (13)
Lymphopenia (Blood and lymphatic system disorders) | 6 (11)
Neutropenia (Blood and lymphatic system disorders) | 17 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 6 (6)
Conjunctivitis (Eye disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 22 (26)
Diarrhoea (Gastrointestinal disorders) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 27 (27)
Nausea (Gastrointestinal disorders) | 43 (67)
Oesophagitis (Gastrointestinal disorders) | 23 (25)
Stomatitis (Gastrointestinal disorders) | 10 (12)
Vomiting (Gastrointestinal disorders) | 11 (15)
Asthenia (General disorders) | 18 (23)
Chest pain (General disorders) | 5 (8)
Fatigue (General disorders) | 14 (16)
Pyrexia (General disorders) | 8 (10)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 10 (10)
Radiation skin injury (Injury, poisoning and procedural complications) | 10 (10)
Haemoglobin decreased (Investigations) | 7 (7)
Neutrophil count decreased (Investigations) | 5 (6)
White blood cell count decreased (Investigations) | 5 (7)
Decreased appetite (Metabolism and nutrition disorders) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Dizziness (Nervous system disorders) | 7 (7)
Dysgeusia (Nervous system disorders) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days